CLINICAL TRIAL: NCT00510614
Title: Tinidazole for Recurrent Bacterial Vaginosis: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mission Pharmacal (Industry)
Responsible Party: Richard H Beigi, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO07030019
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; Recurrent Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Tinidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 1 gram tinidazole twice weekly for 12 weeks
  Interventions: Drug: tinidazole
- B (Placebo Comparator): Placebo twice weekly for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tinidazole — 1 gram twice weekly for 12 weeks
  Other Names: Tindamax
  Arms: A
Drug: Placebo — one pill twice weekly for 12 weeks
  Arms: B

SUMMARY:
This research study is being done to evaluate the use of an oral (by mouth) medication called tinidazole to initially treat BV and then to see if additional treatment with tinidazole keeps women from getting this infection back within 3 months. Tinidazole is currently approved by the United States Food and Drug Administration (FDA) to treat bacterial vaginosis (BV).

This study will evaluate the use of tinidazole to treat a woman's current BV infection and then will look at using tinidazole as a suppressive treatment (taking medication regularly to attempt to decrease the "bad" bacteria from growing back). The suppressive treatment phase will include using tinidazole twice a week compared to using placebo twice a week and then following women for recurrence of BV. The purpose of this study is to determine if tinidazole suppression will prevent BV from coming back within 3 months of treatment.

The investigators hypothesize that women with a history of recurrent bacterial vaginosis who are randomized to a suppressive regimen (a dose of medication given on a regular basis to attempt to control the bacteria that causes bacterial vaginosis) of tinidazole will have lower recurrence rates and a longer time to recurrence of bacterial vaginosis when compared to those women randomized to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 at time of enrollment.
2. Recurrent BV as defined by:

   * 2 previously documented diagnoses of BV in the past 6 months or
   * 3 previously documented diagnoses of BV in the past year
3. Non-pregnant, non-lactating.
4. Premenopausal.
5. Presence of bacterial vaginosis at the enrollment visit using Amsel Criteria (at least 3 of 4):

   * Presence of homogenous vaginal discharge
   * pH of vaginal secretions of > 4.7
   * Presence of a positive "whiff" test of the vaginal secretions upon mixing with 10% KOH
   * Presence of > 20% clue cells on saline microscopy
6. Willingness to undergo randomization to a possible placebo arm (for suppressive therapy).
7. Ability to undergo informed consent.
8. Willingness to refrain from use of any intravaginal products (including douching, contraceptive spermicides, creams, gels, foams).
9. Currently using an acceptable method of birth control (such as a hormonal method including oral contraceptives, Depo Provera, Ortho Evra, abstinence x 60 days, consistent condom use, surgically sterile, lesbian orientation).
10. Willing to refrain from alcohol consumption during use of study medication and three days following completion of medication (which includes the 10 day open label treatment and the entire 3 month suppressive phase of treatment).

Exclusion Criteria:

1. Known active sexually transmitted infection at the time of enrollment with C. trachomatis, N. gonorrhoeae, T. vaginalis, or active (symptomatic) vulvovaginal candidiasis.
2. Current use of anticoagulants/blood thinners (i.e. warfarin, coumadin, heparin).
3. Current use of any of the following medications: lithium, fluorouracil, anticonvulsant/seizure medications, Questran (cholestyramine) or CYP3A4 inducer/inhibitors (i.e. phenobarbital, rifampin, phenytoin, fosphenytoin).
4. Use of Antabuse (disulfiram) currently or within the past 2 weeks.
5. Allergy to metronidazole or tinidazole (related drugs with likely cross-over allergy potential).
6. Use of any antibiotics (oral or vaginal) in the past 7 days.
7. Current use of an IUD, Nuva Ring.
8. Known immunosuppressive condition (i.e. HIV, end-stage renal disease, currently-treated diabetes mellitus, etc.) or on immunosuppressive medications [i.e. steroids, cyclosporine, Protopic (tacrolimus), immunomodulators].
9. Participation in an investigational drug study within the past 30 days.
10. Any condition which in the opinion of the investigator would impose a health risk to the subject or interfere with the evaluation of the study medication or procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Differences in the proportion of women clinically cured at each visit between the two therapy arms will be evaluated using Fisher's-exact test. | at each study visit

SECONDARY OUTCOMES:
Kaplan-Meier product-limit estimation will be used to obtain estimates of the median time to BV recurrence. | at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beigi, MD, MSc., Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States